CLINICAL TRIAL: NCT05580640
Title: Investigating the Efficacy of Osteopathic Manipulative Treatment on Gait Dysfunction Following Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB: 21053
Record Dates: First submitted 2022-09-30; First posted 2022-10-14 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-09

CONDITIONS: Knee Arthroscopy; Knee Arthroplasty; Osteopathic Manipulative Treatment; Gait, Unsteady
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: For this proof-of-concept study we will use a series of case studies. This will allow us to determine if a single session of OMT can improve gait in subjects with prior knee surgery, whether multiple sessions are required to change chronic compensatory musculoskeletal issues, and whether subtle gait anomalies (or improvements), in patients with knee arthroscopy can be detected with the gait analysis system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 months + post knee surgery (Experimental): : For study participation subjects need a history of unilateral knee arthroscopy or arthroplasty performed > 6 months ago with completion of post-operative rehabilitation. Subjects will be between the ages of 21 and 90 years old and the ability to walk for 5-10 minutes on level ground.
  Interventions: Procedure: OMT

INTERVENTIONS:
Procedure: OMT — For this proof-of-concept study we will use a series of case studies. This will allow us to determine if a single session of OMT can improve gait in subjects with prior knee surgery, whether multiple sessions are required to change chronic compensatory musculoskeletal issues, and whether subtle gait anomalies (or improvements), in patients with knee arthroscopy can be detected with the gait analysis system

SUMMARY:
For patients with a history of knee surgery, especially knee arthroplasty, the persistence of abnormal gait kinematics is a frequently encountered issue that can hinder their ability to return to normal daily living.

Muscular imbalances and leg length discrepancy (LLD) following knee arthroplasty can impact a patient's ability to return to a normal gait pattern. In a study of 98 patients who underwent total knee arthroplasty, leg lengthening on the side of the operative knee was reported in 83% of patients as determined by comparing pre- and postoperative leg-length radiographs (Lang JE et al; J. Arthroplasty. 2012;27(3):341-346). LLD can lead to compensations in surrounding joints, muscles, and myofascial structures. Compensatory musculoskeletal changes, including changes in pelvic tilt and curvature of the lumbar spine can alter gait mechanics, lead to mechanical low back pain, and increase the risk of degenerative disc disease (Sheha EDM et al; J. Bone and Joint Surgery, Inc. 2018;6(8)(e6)). In addition, neurologic compensations can occur and include changes in muscular timing and muscular activation patterns. The mainstay of gait rehabilitation following knee surgery is physical therapy (PT) (O'Connor DP et al; J Orthop Sports Phys Ther. 2001;31(7):340-352), where LLD can be addressed with heel lift therapy. The use of Osteopathic Manipulative Treatment (OMT) to address chronic compensatory musculoskeletal changes following knee surgery in order to improve gait has not been extensively studied. Both OMT and PT have been shown to improve gait imbalances in a variety of neurological conditions such as Parkinson's disease, multiple sclerosis, and Prader-Willi syndrome. Previous studies of these neurologic conditions have demonstrated increases in walking velocity, step length, stride length and range of motion of the lower extremities following OMT. It remains to be determined whether OMT can improve gait pattern abnormalities caused by compensatory musculoskeletal patterns that persistent after traditional postoperative knee rehabilitation.

The purpose of this study is to determine if OMT of chronic, compensatory, musculoskeletal issues associated with knee surgery improves gait parameters. In addition to providing objective parameters to assess and validate OMT, future patients recovering from knee surgery might benefit from OMT

DETAILED DESCRIPTION:
Study Design: For this proof-of-concept study we will use a series of case studies. This will allow us to determine if a single session of OMT can improve gait in subjects with prior knee surgery, whether multiple sessions are required to change chronic compensatory musculoskeletal issues, and whether subtle gait anomalies (or improvements), in patients with knee arthroscopy can be detected with the gait analysis system. If the data support our hypothesis, we will request an amendment to the IRB to expand subject numbers and include a control group. Location: MWU Multi-Specialty Clinic Overall Protocol: Informed consent participants will first complete a Knee Outcome Survey, undergo preintervention evaluation of quadriceps strength, knee range of motion, and leg length. Participants will then undergo gait analysis. An Osteopathic physician (KPH) will then diagnose and treat somatic dysfunction.

After OMT, subjects will repeat clinical measures (quadriceps strength, knee ROM, and leg length) and gait analysis to determine the acute effects of OMT. Because chronic compensatory musculoskeletal issues may not be resolved with one session of OMT, subjects will return to the Multi-Specialty Clinic (MSC) for OMT

1x/wk for 2wks. During the fourth week, subjects will repeat the pre-intervention evaluation and gait analysis before and after the fourth and final OMT session. In total, subjects will undergo four gait analysis sessions: two evaluations during the first encounter and two during the fourth week of the study. Detailed protocols for data collection are listed below. Knee Outcome Survey - Activities of Daily Living (KOS-ADL) will be used to measure each subject's current symptoms and functional limitations before and after participation in the study. The KOS-ADL is a

ELIGIBILITY:
Inclusion Criteria:

* Unilateral knee arthroscopy completed > 6 months ago with complete post-operative rehabilitation.
* Able to walk for 5-10 minutes on level ground.

Exclusion Criteria:

* Pregnancy
* Subjects with vestibular impairments or cardiovascular disease
* Inability to walk without the aid of an assistive device (e.g., walker, cane),
* History of neurological disorders including multiple sclerosis, Parkinson's disease or stroke causing gait impairment
* Subjects with additional joint replacements, spinal fusions, or a history of hip, ankle, or foot surgery.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Acute effect of one OMT session on gait | Acute 1hr
  We hypothesize one Osteopathic Manipulative Treatment (OMT) session will increase walking speed and motion efficiency between the operative and non-operative leg in patients with a history of knee surgery. Gait analysis will quantify differences in force and motion, in space and time (spatiotemporal kinetics and kinematics).
Effect of four OMT sessions on gait | 4 weeks
  Patients with knee arthroplasty may have chronic somatic dysfunction that requires several OMT sessions to have an effect. We hypothesize four sessions of Osteopathic Manipulative Treatment (OMT) will increase walking speed and motion efficiency between the operative and non-operative leg in patients with a history of knee surgery. Gait analysis will quantify differences in force and motion, in space and time (spatiotemporal kinetics and kinematics).

CONTACTS AND LOCATIONS:
Locations (1):
- MidwesternU, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No